CLINICAL TRIAL: NCT06488144
Title: A Remotely - Applied Behaviorally- Designed Intervention Incorporating Gamification, Social Incentives, and Health Coaching to Improve Durability of Physical Therapy for Knee Osteoarthritis (ReAKTIV)
Brief Title: Rehabilitation for Arthritis of The Knee: mainTaining Improvement for Veterans
Acronym: ReAKTIV
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: F4770-R; RX004770 (Other Grant/Funding Number: VA Rehabilitation Research & Development)
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee
Keywords: physical therapy; health coach; behavioral intervention
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No Intervention (No Intervention): Neither Intervention
- Health Coaching, No Incentives (Experimental): Receives a Health Coach but no Incentive Program
  Interventions: Behavioral: Health coach
- No Health Coach, Receives Incentives (Experimental): Does not receive a health coach but does receive the incentive program.
  Interventions: Behavioral: Remote Incentive Program
- Health Coaching, Receives Incentives (Experimental): Receives both a health coach and the incentive program
  Interventions: Behavioral: Health coach; Behavioral: Remote Incentive Program

INTERVENTIONS:
Behavioral: Health coach — Health Coaching
  Arms: Health Coaching, No Incentives; Health Coaching, Receives Incentives
Behavioral: Remote Incentive Program — Behavioral incentive program including gamification, social incentivization, and monitoring.
  Arms: Health Coaching, Receives Incentives; No Health Coach, Receives Incentives

SUMMARY:
The aims are to determine whether 1) an incentive based on behaviorally-enhanced gamification and social incentives and 2) health coaching can promote adherence to exercise and physical activity after physical therapy for osteoarthritis of the knee (KOA). The research design is a randomized clinical trial with factorial design

This randomized clinical trial of 254 patients using a factorial design will leverage a clinical trial platform developed through the University of Pennsylvania that allows for the remotely capture important patient-reported outcomes and other interaction through a participant's smart phone. The investigators will randomize participants to receive social incentives with gamification to promote adherence to prescribed exercises as well as maintenance of greater levels of physical activity and compare to controls that receive a Fitbit but no additional incentive. Participants may also be randomized to receive a health coach. The investigators will utilize mobile applications for smart phones and wearable activity trackers through the Way-to-Health platform and assess, in real time, the impact of the interventions on patient-reported function and pain (as measured by the Knee Osteoarthritis Outcome Score) as well as physical activity. Participants will be followed for 2 years, with a total of 5 in-person visits.

Knee osteoarthritis (KOA) is one of the most prevalent and disabling conditions among Veterans and accounts for high morbidity and high costs for the VA. Importantly, while physical therapy is valuable for patients with KOA, lack of adherence to home exercises and low overall physical activity limit the durability of response. The current proposal aims to address two important knowledge gaps in the management of KOA in order to improve pain and function.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a high-priority problem among the aging population, and in particular, among Veterans. Few interventions have been shown effective in the long-term management of symptoms. Current guidelines for non-operative KOA management include strong recommendations for exercise delivered through standard physical therapy (PT) and the promotion of greater physical activity. Standard physical therapy (PT) interventions characterized by 6-8 week of supervised exercises (e.g., strengthening peri-articular tissues) and mobility training (e.g., improving biomechanics and movement patterns) are safe and effective at improving and facilitating mobility, activity participation, and overall quality of life. While PT is a recognized and necessary aspect of KOA care, its clinical benefits are often short-lived and begin to decline following PT due to poor long-term adherence - leading physicians to increasingly rely on the use of non-steroidal anti-inflammatories and opioids over time. The lack of effective strategies to sustain the clinical benefits achieved in PT for individuals with KOA remains a critical gap.

The investigators aim to study two interventions designed based on their ability to address 5 key theories for maintaining behaviors that are supported by the literature. Specifically, the proposed study will evaluate a remote and behaviorally-designed intervention in combination with health coaching to influence long-term behavioral change after standard-of-care PT. The behavioral intervention utilizes tools such as goal setting, gamification (the use of game design elements), loss aversion, monitoring, and social incentives, to 1) increase motivation, 2) improve self-monitoring and self-regulation, 3) provide psychological and physical resources, 4) influence the development of healthy long-term habits, and 5) a provide supportive environment with social support. The behavioral intervention will be studied combined with health coaching with a focus on the same goals but through motivational interviewing to address personal, environmental, and social barriers. The investigators aim to clearly quantify the value of each as well as their value when used in combination.

The investigators has already utilized concepts from behavioral economics (a scientific field aiming to understand how to motivate individuals) to develop remotely-applied interventions that incorporate the concepts of gamification, social incentives, and loss aversion to promote improvements in physical activity using an innovative web-based platform. The investigators SPiRE-funded pilot study "Marching On for Veterans with Osteoarthritis of the Knee" demonstrated excellent feasibility, rapid recruitment, improvements in reported symptoms, and high patient satisfaction. The multi-site study is actively enrolling Veterans and is ahead of schedule.

The investigators propose to fill important knowledge gaps in this area with a large, pragmatic clinical trial. In this study, the investigators will randomize in a factorial design to receive no intervention, the remote behavioral intervention, a remote health coach, or both, after being released from a standard PT intervention with proven efficacy in order to promote the maintenance of symptomatic gains observed during PT. To accomplish these aims, the investigators will utilize innovative mobile applications for smart phones through the Way-to-Health (WTH) platform and assess, in real time, the impact of the intervention on the primary outcome of patient-reported symptoms as measured by the Knee Osteoarthritis Outcome score. The investigators will also monitor adherence to specific knee-related exercises at home. Way to Health allows for the recording of outcomes in real time, as they occur, thereby avoiding information bias due to poor recall and participation bias. The investigative team includes investigators with experience conducting similar trials using this infrastructure as well as expertise in behavioral economics and motivational interviewing. The study also involves a centralized organizational structure in close collaboration with investigators across the country.

Aim 1: To determine if a personalized and remotely-applied behavioral intervention based on insights from behavioral economics can sustain the symptomatic gains following physical therapy for KOA. Hypothesis: A remotely-applied program will result in maintenance of higher KOOS scores after PT by promoting greater adherence, self-efficacy, habituation, and social support.

Aim 2: To determine if a remote health coach can sustain the symptomatic gains following physical therapy for KOA. Hypothesis: Those that are randomized to receive a health coach will maintain higher KOOS scores after PT.

Aim 3: To determine how the behavioral intervention and health coaching interventions interact with each other. Hypothesis: The effect of both interventions will be additive such that the greatest improvement in symptoms will occur among those that receive both interventions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis or chronic knee osteoarthritis.
* Age between 40-90 years
* Initiating physical therapy for KOA (has initial appointment within the next month or had first PT visit within the last 7 days)
* To be randomized: PT feels that they are able to safely and reliably participate in ongoing exercise.
* To be randomized: must have completed at least 4 virtual or in-person appointments with PT
* To be randomized: must sync their Fitbit at least monthly.

Exclusion Criteria:

* Lack of a smart phone allowing interaction with the WTH platform
* Inability to walk 2 blocks without assistance
* Poorly controlled crystalline arthritis or other diagnosis of inflammatory arthritis.
* Treating provider or LSI believes life-expectancy is <1 year
* Based on LSI or treating provider discretion: exclusions may occur for severe heart failure, unstable angina, end stage renal disease, severe chronic obstructive or other pulmonary disease, or other chronic illness felt to limit participants ability to participate in exercise or resulting in potential safety risk
* Severe pain in a non-knee area limiting daily function
* Non-English speakers or poor reading ability limiting ability to interact with text messages.
* Pregnancy
* Receiving physical therapy outside of the VA.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
KOOS (Knee Osteoarthritis Outcome Score) | all available measures between 6-18 months (time-averaged effect)
  The KOOS score is a validated and widely used measure of knee-related pain and physical functioning that has been validated in both knee injury and KOA populations. The KOOS measures symptoms and disability on five subscales: Pain, other Symptoms, Function in Activities of Daily Living, Function in Sports and Recreation, and Quality of Life (QOL). Range is from 0-100 for each subscale with lower scores suggesting worse patient experience.

SECONDARY OUTCOMES:
Average Daily Step Counts | 0-18 Months
  Change in average daily step counts (averaged over the prior month) throughout follow-up (time-averaged effect).
Change in Self Efficacy for excercise | 6-18 months
  Self-efficacy for exercise scale (change from baseline; time-averaged effect). Range 0-100 with higher scores representing more confidence in exercise.
Change in gait speed | 6-18 months
  Change in walking speed over a 4 meter testing zone (time-averaged effect)
30 second sit-to-stand | 6-18 months
  Number of times a person can stand and sit within 30 seconds (time-averaged effect)
Patient Reported Outcomes Measurement Information System Pain Intensity | 6-18 Months
  Change from baseline in PROMIS Pain Intensity (time-averaged effect). Scale 0-100 (higher score indicates more pain).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua F. Baker, MD MSCE, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (5):
- United States (5):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No